CLINICAL TRIAL: NCT05648305
Title: Root Canal Treatment is a Common Intervention for Military Patients Suffering From- or at Risk of Suffering From- Endodontic Disease. This Retrospective Cohort Study Assesses the Influence of (a) Root Canal Complexity Using the Restorative Index of Treatment Need (RIOTN) Index and (b) Operator Skill (Clinicians Who Had Received Additional Post-graduate Root Canal Treatment Training, on Survival (Tooth Present at End of Study Period) and Success (Radiographic Apical Healing) of Root Canal Treatment
Brief Title: The Influences of Root Canal Complexity and Clinician Training on Root Canal Treatment Outcomes.
Status: Completed | Type: Observational
Sponsor: Defence Primary Health Care, UK (Other Government)
Collaborators: Eastman Dental Insitute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DefencePHC
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Root Canal Infection
Keywords: Root Canal Treatment
MeSH Terms: interventions — Dental Implantation, Endosseous, Endodontic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Dental Practitioners: Cohort 1 consisted UK Armed Forces Personnel that received root canal treatment within the study period by General Dental Practitioners.
  Interventions: Procedure: Root Canal Treatment/ Re-treatment
- Dentists with Specialist Interest (DWSI): Cohort 2 consisted UK Armed Forces Personnel that received root canal treatment within the study period by DWSI, clinicians that had undertaken a 1-year post-graduate programme in Endodontics.
  Interventions: Procedure: Root Canal Treatment/ Re-treatment

INTERVENTIONS:
Procedure: Root Canal Treatment/ Re-treatment — The provision of Root Canal Treatment for teeth with Endodontic infection or to prevent Endodontic infection.
  Other Names: Endodontic Therapy

SUMMARY:
This is an observational study that assess the impacts of (a) root canal treatment complexity and (b) clinical training on (1) root canal treatment success and (2) tooth survival, in a United Kingdom Armed Forces cohort.

DETAILED DESCRIPTION:
Background and Study Aims. This observational cohort study evaluates root canal treatment outcomes, using survival and success as the outcome measures. It aims to assess the influence of operator skill and RIOTN complexity on the clinical outcomes of RCT procedures previously undertaken within the UK Armed Forces.

Participation UK Armed Forces personnel that had previously received root canal treatment between 01/01/2015 and 01/09/2020.

Method

A Defence Statistics programme was used to identify cohorts of patients treated for Endodontic disease by GDPs and DWSI (GDPs who had undertaken a 1 year post-graduate training programme in Endodontics). The researcher group was calibrated to the study's method and this was initially piloted on 5 patient records, with further calibration undertaken until researcher consistency was achieved via inter-operator reliability testing. The researchers subsequently reviewed 1600 patient records, eventually establishing a cohort of 1267 patients (580 - Group 1 (GDP) and 687 - Group 2 (DWSI). The clinical records and radiographs of these groups were reviewed for the following:

1. Tooth survival 2. RIOTN complexity at the time of treatment 3. RCT success (apical healing). Secondary factors assessed included: age, gender, smoking status, diabetic status, steroid status, presence of an indirect restoration, presence of a post, reasons for tooth loss (if tooth did not survive).

The collection of data has now been completed and is ready for analysis.

Risks and Benefits This study will benefit Defence Primary HealthCare and UKAF personnel as it will influence and shape future care provision for Endodontic disease within the military. There are no identified risks of participation.

Study Location The study is being run from the Defence Centre for Rehabilitative Dentistry, Evelyn Woods Road, Aldershot, GU11 2LS. The study is evaluation the outcomes of clinical practitioners working within the 200+ Dental Centres within the UK and overseas locations.

Funding There is no established funding for this study. There are no commercial or other conflicts of interest.

ELIGIBILITY:
Inclusion Criteria:

* Served/ were serving within the UK Armed Forces.
* Male and female.
* Physically able to tolerate root canal treatment/ re-treatment procedures.
* Received root canal treatment/ re-treatment for Endodontic disease by either a GDP or Dentist with Specialist interest (DWSI).
* Aged between 18 - 70..
* 12-month (or longer) post root canal treatment review radiograph and consultation.
* Smoking and non-smoking patients
* With and without Diabetes Mellitus 2
* Taking/ not-taking steroid medications
* With/ without other medical conditions.

Exclusion Criteria:

* On longer serving in the military within 12-months of root canal treatment completion.
* Unable to tolerate root canal treatment/ re-treatment
* No clinical follow-up of tooth (survival).
* No radiographic follow-up of tooth (success).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and Female personnel serving within the UK Armed Forces that had received root canal treatment during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 1267 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
1. Tooth survival | 6-months - 48-months post-treatment.
  Tooth still present in the mouth at end of trial period.
2. Root Canal Treatment Success | 6-months - 48-months post-treatment.
  The absence of signs, symptoms and evidence of radiographic peri-apical radiolucency resolution.

CONTACTS AND LOCATIONS:
Overall Officials: Neil MacBeth, BDS PhD, Study Chair — Defence Primary Healthcare

IPD SHARING:
Plan to Share IPD: No
The data belongs to the UKAF. Requests for data sharing would require MOD approval.